CLINICAL TRIAL: NCT07379034
Title: The Effect of ShotBlocker and Vibration Pen on Pain During Vaccination in Healthy Infants: A Randomized Controlled Study
Brief Title: The Effect of ShotBlocker and Vibration on Pain During Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Sümeyye EKİCİ, Research Assistant, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Research1
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Vaccination; Pain; Infant; Shotblocker; Vibration
Keywords: vaccination; pain; infant; Shotblocker; Vibration
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental 1 (Experimental): ShotBlocker Group
  Interventions: Other: ShotBlocker Group
- Experimental 2 (Experimental): Vibration device group
  Interventions: Other: Vibration Group
- Control (No Intervention): Routine nursing care

INTERVENTIONS:
Other: ShotBlocker Group — ShotBlocker is a plastic medical device with multiple blunt projections that is applied by pressing on the skin during injection. It aims to reduce pain transmission through activation of the Gate Control Theory by stimulating multiple sensory nerve endings and diverting the infant's attention from the painful stimulus.
  Arms: Experimental 1
Other: Vibration Group — The vibration pen is a battery-operated device that delivers high-frequency mechanical vibrations and is applied near the injection site. It aims to reduce perceived pain intensity by stimulating large-diameter nerve fibers and inhibiting pain transmission at the "gate" level.
  Arms: Experimental 2

SUMMARY:
This study was conducted to investigate the effects of ShotBlocker and a vibration pen on pain in infants during routine vaccination. In this randomized controlled trial, 96 healthy infants aged 2-6 months were included. The infants were randomized into three groups: vibration pen, ShotBlocker, and control. Pain was assessed before, during, and after the procedure using the FLACC scale.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infant aged 2-6 months
* Written consent from the parent

Exclusion Criteria:

* Premature infants born before 37 weeks
* Infants with severe neurodevelopmental disorders
* Presence of acute infection or fever
* History of a previous serious vaccine reaction

Ages: 2 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-01-23 (Actual); Study Completion 2026-01-23 (Actual)

PRIMARY OUTCOMES:
FLACC Scale | up to 6 months
  The FLACC score will be used as the data collection tool. The FLACC scale is a valid and reliable measure that assesses infant pain by evaluating five domains-facial expression, leg movement, activity level, crying, and consolability-and scores pain on a scale from 0 to 10.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Yakutiye, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No